CLINICAL TRIAL: NCT01252901
Title: Registry for Patients With WT1 Mutation Associated Diseases
Brief Title: Registry for Patients With Wilms' Tumor Suppressor Gene 1 (WT1) Mutation Associated Diseases
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: WT1 Registry
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Denys-Drash Syndrome; Frasier Syndrome; Nephrotic Syndrome; Wilms Tumor
Keywords: WT1; Wilms Tumor; Denys-Drash Syndrome; Nephrotic Syndrome; Proteinuria
MeSH Terms: conditions — Denys-Drash Syndrome; Frasier Syndrome; Nephrotic Syndrome; Wilms Tumor; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Wilms' tumor suppressor gene 1 (WT1) encodes for a transcription factor which plays an important role during urogenital development. Patients carrying a WT1 germline mutation show symptoms like proteinuria, Wilms tumors, genital malformations and kidney failure. Milder variants are possible and classification is not always possible. In this registry we are collecting detailed clinical data of affected individuals to establish genotype-phenotype correlations with the greater goal to optimize patient care.

DETAILED DESCRIPTION:
The Wilms' tumor suppressor gene 1 (WT1) encodes for a transcription factor which plays an important role during urogenital development. Patients carrying a WT1 germline mutation show symptoms like proteinuria, Wilms tumors, genital malformations and kidney failure, which usually occur in early childhood. Milder variants are possible and classification as one of the three rare syndromes associated with WT1 mutations (Denys-Drash syndrome, Frasier syndrome or WAGR syndrome) is not always possible. In this registry we are collecting detailed clinical data of affected individuals to establish genotype-phenotype correlations with the greater goal to optimize patient care.

ELIGIBILITY:
Inclusion Criteria:

* Germline mutation in WT1 gene

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with WT1 mutation
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2010-10; Primary Completion 2013-11 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Lehnhardt, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätskrankenhaus Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Background] Royer-Pokora B, Beier M, Henzler M, Alam R, Schumacher V, Weirich A, Huff V. Twenty-four new cases of WT1 germline mutations and review of the literature: genotype/phenotype correlations for Wilms tumor development. Am J Med Genet A. 2004 Jun 15;127A(3):249-57. doi: 10.1002/ajmg.a.30015. PMID 15150775
- [Background] Mucha B, Ozaltin F, Hinkes BG, Hasselbacher K, Ruf RG, Schultheiss M, Hangan D, Hoskins BE, Everding AS, Bogdanovic R, Seeman T, Hoppe B, Hildebrandt F; Members of the APN Study Group. Mutations in the Wilms' tumor 1 gene cause isolated steroid resistant nephrotic syndrome and occur in exons 8 and 9. Pediatr Res. 2006 Feb;59(2):325-31. doi: 10.1203/01.pdr.0000196717.94518.f0. PMID 16439601
- [Background] Ruf RG, Schultheiss M, Lichtenberger A, Karle SM, Zalewski I, Mucha B, Everding AS, Neuhaus T, Patzer L, Plank C, Haas JP, Ozaltin F, Imm A, Fuchshuber A, Bakkaloglu A, Hildebrandt F; APN Study Group. Prevalence of WT1 mutations in a large cohort of patients with steroid-resistant and steroid-sensitive nephrotic syndrome. Kidney Int. 2004 Aug;66(2):564-70. doi: 10.1111/j.1523-1755.2004.00775.x. PMID 15253707
- [Background] Kist-van Holthe JE, Ho PL, Stablein D, Harmon WE, Baum MA. Outcome of renal transplantation for Wilms' tumor and Denys-Drash syndrome: a report of the North American Pediatric Renal Transplant Cooperative Study. Pediatr Transplant. 2005 Jun;9(3):305-10. doi: 10.1111/j.1399-3046.2005.00311.x. PMID 15910385
- [Background] Aucella F, Bisceglia L, De Bonis P, Gigante M, Caridi G, Barbano G, Mattioli G, Perfumo F, Gesualdo L, Ghiggeri GM. WT1 mutations in nephrotic syndrome revisited. High prevalence in young girls, associations and renal phenotypes. Pediatr Nephrol. 2006 Oct;21(10):1393-8. doi: 10.1007/s00467-006-0225-0. Epub 2006 Aug 15. PMID 16909243
- [Background] Chesney RW. Why is the oncogene WT1 in the developing kidney and what is it doing there? Pediatr Nephrol. 2002 Dec;17(12):990-2. doi: 10.1007/s00467-002-0927-x. Epub 2002 Oct 1. No abstract available. PMID 12520325
- [Background] Klamt B, Koziell A, Poulat F, Wieacker P, Scambler P, Berta P, Gessler M. Frasier syndrome is caused by defective alternative splicing of WT1 leading to an altered ratio of WT1 +/-KTS splice isoforms. Hum Mol Genet. 1998 Apr;7(4):709-14. doi: 10.1093/hmg/7.4.709. PMID 9499425
- [Background] Pelletier J, Bruening W, Kashtan CE, Mauer SM, Manivel JC, Striegel JE, Houghton DC, Junien C, Habib R, Fouser L, et al. Germline mutations in the Wilms' tumor suppressor gene are associated with abnormal urogenital development in Denys-Drash syndrome. Cell. 1991 Oct 18;67(2):437-47. doi: 10.1016/0092-8674(91)90194-4. PMID 1655284
- See also: University Medical Center Hamburg-Eppendorf — http://www.uke.de
- See also: Gesellschaft für Pädiatrische Nephrologie — http://www.gp-nephrologie.de
- See also: DSD Network for Disorders of Sex Development — http://www.netzwerk-is.de/
- See also: Das Informationsportal der Gesellschaft für Pädiatrische Onkologie und Hämatologie — http://www.kinderkrebsinfo.de